CLINICAL TRIAL: NCT00268515
Title: Aerosol Cyclosporine for Prevention of Lung Rejection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: 349; R01HL059490 (NIH)
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-12

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Cyclosporine; Tacrolimus; Prednisone; Azathioprine

INTERVENTIONS:
Drug: cyclosporine
Drug: tacrolimus
Drug: prednisone
Drug: azathioprine

SUMMARY:
To evaluate the efficacy of aerosolized cyclosporine given in addition to the standard oral immunosuppressive drug regimen, in preventing acute rejection immediately after lung transplantation

DETAILED DESCRIPTION:
BACKGROUND:

Success with lung transplantation has largely been due to the introduction of cyclosporine which has proved effective in controlling lung allograft rejection. Nevertheless, acute and chronic rejection are prevalent in spite of immunosuppressive drug regimens based on oral cyclosporine. In fact, rejection is more common in recipients of lung allografts than those who receive other solid organs. Acute rejection is treated with pulsed methylprednisolone and anti-lymphocyte globulin and consequently recipients are subject to increased risk of infection and drug toxicity. The hypothesis tested in the study was that delivery of cyclosporine to the transplanted lung by aerosol inhalation would achieve higher concentrations of cyclosporine in the graft than when it was delivered via the bloodstream and that higher concentrations in the graft would prevent rejection more effectively than systemic immune suppression with the same or reduced toxicity.

Cellular rejection occured in over 90% of the patients within the first year and often progressed to obliterative bronchiolitis (OB) which was the most common cause of death one year after transplant. In 1988, the lung transplant group at the University of Pittsburgh decided to pursue cyclosporine aerosol for the treatment for acute rejection. After animal testing, initial human experiments were performed, which suggested that cyclosporine aerosol decreased the prevalence of acute rejection and the development of obliterative bronchiolitis.

DESIGN NARRATIVE:

This prospective double blind randomized trial was designed to evaluate the efficacy of cyclosporine aerosol versus placebo aerosol as an adjuvant to oral immunosuppression with tacrolimus, prednisone, and azathioprine. The hypotheses tested included: 1) acute rejection would be lower in the patients receiving cyclosporine aerosol, 2) maintenance cyclosporine aerosol would result in reduced incidence of OB, 3) cytokines and chemokine release would be suppressed, 4) patients receiving cyclosporine aerosol would require less systemic immunosuppression and 5) there would be a lower incidence of opportunistic and bacterial infections as a consequence of more effective immunosuppressive therapy. Another specific aim of the study was to determine the optimal dose of cyclosporine aerosol that reduced rejection and/or OB and to correlate radioisotopically labeled inhalation studies with more easily measurable indices that affected the deposition of aerosolized medications.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-04; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Iacono — University of Pittsburgh

REFERENCES:
- [Background] Burkart GJ, Smaldone GC, Eldon MA, Venkataramanan R, Dauber J, Zeevi A, McCurry K, McKaveney TP, Corcoran TE, Griffith BP, Iacono AT. Lung deposition and pharmacokinetics of cyclosporine after aerosolization in lung transplant patients. Pharm Res. 2003 Feb;20(2):252-6. doi: 10.1023/a:1022275222207. PMID 12636164
- [Result] Iacono AT, Johnson BA, Grgurich WF, Youssef JG, Corcoran TE, Seiler DA, Dauber JH, Smaldone GC, Zeevi A, Yousem SA, Fung JJ, Burckart GJ, McCurry KR, Griffith BP. A randomized trial of inhaled cyclosporine in lung-transplant recipients. N Engl J Med. 2006 Jan 12;354(2):141-50. doi: 10.1056/NEJMoa043204. PMID 16407509